CLINICAL TRIAL: NCT03077009
Title: Functional Improvement and Ultrasound Tissue Characterisation of the Achilles Tendon Following Sodium Hyaluronate Injection for Plantaris Friction Syndrome
Brief Title: Functional Improvement and UTC of the Achilles Tendon After Sodium Hyaluronate Injection for Plantaris Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fortius Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FortiusClinic
Record Dates: First submitted 2017-02-12; First posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-02

CONDITIONS: Plantaris Friction Syndrome; Non-Insertional Achilles Tendinopathy
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Patients with confirmed plantaris friction syndrome will be offered hyaluronic acid injection into the space between the Plantaris and Achilles tendons
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Drug: Hyaluronic Acid — Ultrasound guided injection for plantaris friction syndrome
  Other Names: Ostenil

SUMMARY:
This is a study to assess the benefit of sodium hyaluronate (Ostenil) injection for plantaris friction syndrome (PFS) associated with midportion Achilles tendinopathy. Functional outcome scores will be recorded prior to treatment and at regular intervals up to 2 years. Changes in tendon structure will be assessed using ultrasonographic tissue characterisation (UTC). UTC will be performed prior to treatment and also at regular intervals up to 6 months following injection.

DETAILED DESCRIPTION:
Introduction Midportion Achilles tendinopathy is a common source of disability, with typical features including pain, swelling and dysfunction [Roche]. The causes are multifactorial [Roche]. First line treatment is typically non operative and includes an eccentric loading program [Alfredson-1998], high volume injection [Chan], platelet rich plasma [de Vos JAMA 2010], sclerosing agent injections [Alfredson-2005] , shock wave therapy [Lynen][Saxena] and for resistant cases, surgery [Alfredson-2011].

Plantaris friction syndrome (PFS) One possible cause of midportion Achilles tendinopathy is plantaris friction syndrome (PFS). In this subset of patients, the pain is located to the postero-medial aspect of the Achilles tendon. The plantaris tendon is a small vestigial tendon originating from the lateral femoral condyle, crossing obliquely to the medial side of the Achilles tendon and inserting into the medial side of the calcaneum. The anatomy at the insertion is highly variable. Over 80% of plantaris tendons insert separately to the Achilles tendon [Daseler]. Biomechanical evidence suggests that the plantaris tendon is stiffer and stronger than the Achilles tendon [Lintz]. Under load therefore, differential movement between the tendons may occur. Subsequently the plantaris tendon can become tendinopathic and thickened. Adhesions may develop between it and the adjacent Achilles tendon [Bedi], initiating medial midportion Achilles tendinopathy. Sensitization of the nerve endings in the fat layer between the Achilles and plantaris has also been demonstrated. The optimal treatment of PFS is currently unclear. Treatments include physiotherapy, injection and surgical excision [Bedi][Pearce][Weinberg][Calder-2014][Alfredson-2011].

Sodium Hyaluronate One potential treatment is injection with sodium hyaluronate which is a viscosupplement solution. It has primarily been used for joint lubrication in arthropathy, but can also be used for tendinopathy [Lynen]. Ostenil Tendon is a sodium hyaluronate solution that potentially acts in several ways to reduce pain. One mode is to act as a lubricant between tendons or between the tendon and its sheath [Akasaka 2005][Akasaka 2006][Nishida][Kumar][St Onge]. It may also promote tendon healing [Chen][Yagishta]. According to unpublished work, Ostenil Tendon significantly reduced pain at 6 weeks for peroneal and also midportion Achilles tendinopathy [Company literature]. It may also act as a medium to allow free passage of nutrients to the tendon [Hagberg]. Sodium hyaluronate injection placed in the interval between the plantaris tendon and Achilles tendon could potentially reduce friction and subsequently pain. Although the effect of sodium hyaluronate injections have been reported in the hip and knee, no previous studies have reported its efficacy for PFS. The primary aim of the current study is to assess the impact of sodium hyaluronate injections in patients with PFS.

Ultrasound tissue characterization Methods of assessing the Achilles tendon for tendinopathy continue to be debated. Common methods include ultrasound and magnetic resonance imaging [Khan][Astrom]. A novel assessment tool is ultrasound tissue characterization (UTC) which uses ultrasound to quantify tendon structure [van Schie][Docking-2015][Docking-2016][Rosengarten][Bedi].

Structural integrity of the tendon matrix is categorized in four echo types (1-green, 2-blue, 3-red, 4-black). Echo types 1 and 2 reflect aligned fibrillar structure, whereas types 3 and 4 indicate disorganised tissue [Bedi]. The entire length of the tendon can be analyzed with a minimum detectable difference in structure to be 1% [Docking-2015]. Bedi et al showed significant improvement in UTC following excision of plantaris for midportion Achilles tendinopathy [Bedi]. However this study was limited because UTC images were not performed at a uniform time pre- and post- surgery [Bedi]. Masci et al found improvement in UTC echo-structure at 6 month follow-up post plantaris excision combined with improvement in VISA-A scores [Masci]. It is debated as to whether fibrillar integrity and matrix organisation correlate with symptoms. For example, a study in elite Australian football players showed that UTC changed following pre-season training, but all players remained asymptomatic at the start and end of the study [Rosengarten]. Ultrasound studies have also questioned the relationship of tendon structure in tendinopathy and patient function [Khan][McAuliffe]. In a study of gymnasts, clinical assessment has only moderate correlation with ultrasound and MR appearances [Emerson].

Given the novelty of UTC for the Achilles tendon, the secondary aim of this study is to assess whether UTC changes following treatment for PFS and to correlate any changes with functional outcome scores.

Aims summary

1. To determine changes in Achilles tendon matrix structure using UTC before and after treatment (6 month follow up)
2. To assess medium term (2 years) effectiveness of a sodium hyaluronate injection in the space between the plantaris and Achilles tendons for midportion Achilles tendinopathy which is associated with PFS.
3. To correlate UTC changes with functional scores

Hypothesis The alternate hypotheses are that sodium hyaluronate injection improves both 1) function and 2) structure of the Achilles tendon for PFS.

Outcome measures

* Ultrasonographic tissue characterisation (UTC)
* Functional scores - Victorian Institute of Sports Assessment-Achilles (VISA-A) [Robinson] and Foot and Ankle Outcome scores (FAOS)

Methods This will be a single centre prospective case series of patients in whom PFS has been diagnosed based upon clinical examination by a Consultant foot & ankle surgeon, physiotherapist and imaging. Patients will be prospectively followed up with pre and post intervention patient reported outcome scores.

Sample Population 33 patients diagnosed with PFS will be identified and invited to participate in the study once the decision has been made to treat with sodium hyaluronate.

Inclusion Criteria Patients aged 18-75 years Able to provide informed consent Diagnosis of PFS requiring sodium hyaluronate injection Able to follow physiotherapy instructions Exclusion Criteria Previous Achilles tendon surgery Previous injection therapy for Achilles midportion tendinopathy Age < 18 >75 years Active local infection Active bleeding disorder or anticoagulant therapy Allergies to lignocaine or sodium hyaluronate Active deep vein thrombosis

Patient Recruitment and Consent All patients will be given the information sheet regarding the study and will be consented by the CI or the Fortius foot and ankle fellow. All be patients will be recruited and treated at the Fortius Clinic.

Proposed treatment will include one or two sodium hyaluronate (Ostenil Tendon) injections. Physiotherapy is a routine part of current treatment, usually provided off site.

Injection protocol All injections will be carried out by a Consultant Radiologist at the Fortius Clinic. Approximately 3-5mm of 1% lignocaine will be injected to create a plane between Plantaris and the medial Achilles tendon. Subsequently, 2-3ml of Ostenil Tendon (sodium hyaluronate) will be injected into the space between the Achilles and plantaris tendons.

UTC assessment UTC assessment at 6 and 12 weeks is a routine part of our current treatment protocol for PFS and allows guidance of treatment. Patients will have pre and post treatment UTC assessment of the Achilles tendon. For the purposes of the study, an extra UTC assessment will be performed at 6 months, during part of their routine clinical follow up appointment. This final UTC assessment will be provided free to the patients. All UTC assessments will be conducted by the same experienced physiotherapist.

Follow up Patient reported outcome scores will be completed prior to treatment and at 6 weeks, 3 months,6 months, 1 and 2 years. Outcome scores at 1 and 2 years will be performed online via an automated email system.

UTC will be conducted at 6 weeks, 3 months and 6 months.

Ethical Issues:

Patients will be free to choose to participate or not in the study. If they choose not to participate it will not affect their treatment in any way.

No patient or volunteer will take part in the study without giving written informed consent and we will exclude those patients who are unable to give this consent.

Legal Issues:

There are no legal issues identified that will affect this study.

Management issues:

This study will take place at the Fortius Clinic, which is a private clinic. The patients included would be receiving one or two sodium hyaluronate injections, and two UTC assessments as part of the routine treatment of PFS. They will be charged for this as normal. There will be no additional charge for the final UTC assessment at 6 months.

Risks:

Patients agreeing to take part in the study will be receiving the routine treatment for PFS that they would be receiving even if the study was not taking place. There are therefore no additional risks to the patient.

Data collection All data collection will be done within the premises of the Fortius clinic by members of the clinical team, which includes a physiotherapist who works on site for the Tendon Performance Clinic. In addition to the outcome score and UTC data information regarding patient demographics, medical history and treatment will also be collected.

Data confidentiality Data will be stored in Fortius/Tendon Performance Clinic computers which are password protected and comply with information governance guidelines. No one outside the clinical team will have access to the data.

Any information that leaves the clinic will have patient identifiable information removed. All of the results will be analysed and published using anonymous data only. Details about patient's involvement in the study will also be recorded in patients' medical records held by the Fortius Clinic/Tendon Performance Clinic.

Power analysis In 18 asymptomatic elite Australian football players, UTC demonstrated improvement in Achilles tendon structure over a 5 month period following pre-season training [Docking-2016]. Bedi et al reported UTC changes following Plantaris excision and ventral paratendinous Achilles tendon scraping in athletes. In 11 patients, the fibrillar structure of the Achilles tendon improved from 90 to 96%, SD 8% p=.04. Mean VISA-A scores improved from 51 to 95, SD 12, p=.0001. Regarding sodium hyaluronate injection, only one study was found assessing its use for midportion Achilles tendinopathy [Lynen]. Lynen et al compared two paratendinous injections with three ESWT treatments given at weekly intervals in 62 patients. No previous studies have assessed its use for PFS.

Considering the limited evidence available, we estimate the sample size required to demonstrate improvements in UTC (assuming change in type 1 and 2 echo types from 90% to 96%, SD 8%) to be at least 28 patients. With an expected drop out rate of 15%, we plan to recruit 33 patients to the study.

Statistical analysis Analyses will be conducted using a statistical package. A paired t test will be used to compare pre and post treatment VISA-A scores. UTC results will be compared using Wilcoxon signed rank test (non parametric data). A p value of 0.05 will be defined as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years
* Able to provide informed consent
* Diagnosis of PFS requiring sodium hyaluronate injection
* Able to follow physiotherapy instructions

Exclusion Criteria:

* Previous Achilles tendon surgery
* Previous injection therapy for Achilles midportion tendinopathy
* Age < 18 >75 years
* Active local infection
* Active bleeding disorder or anticoagulant therapy
* Allergies to lignocaine or sodium hyaluronate
* Active deep vein thrombosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2017-03-20 (Estimated); Primary Completion 2020-03-20 (Estimated); Study Completion 2020-03-20 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Tissue Characterisation (UTC) | up to 6 months post intervention
  Structural assessment of the Achilles tendon using ultrasound

SECONDARY OUTCOMES:
Foot and Ankle Outcome Score (FAOS) Functional outcome | up to 2 years post intervention
  Validated patient questionnaire to assess pain, quality of life and activities of daily living. To be competed via email or on site when attending clinical appointments
Victorian Institute of Sports Assessment-Achilles (VISA-A) | up to 2 years post intervention
  Validated patient questionnaire to measure disability caused by Achilles tendon symptoms. To be competed via email or on site when attending clinical appointments

CONTACTS AND LOCATIONS:
Overall Officials: James Calder, MD FRCS, Principal Investigator — Fortius Clinic, London
Locations (1):
- Fortius Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] St Onge R, Weiss C, Denlinger JL, Balazs EA. A preliminary assessment of Na-hyaluronate injection into "no man's land" for primary flexor tendon repair. Clin Orthop Relat Res. 1980 Jan-Feb;(146):269-75. PMID 6768485
- [Background] Chen WY, Abatangelo G. Functions of hyaluronan in wound repair. Wound Repair Regen. 1999 Mar-Apr;7(2):79-89. doi: 10.1046/j.1524-475x.1999.00079.x. PMID 10231509
- [Background] Yagishita K, Sekiya I, Sakaguchi Y, Shinomiya K, Muneta T. The effect of hyaluronan on tendon healing in rabbits. Arthroscopy. 2005 Nov;21(11):1330-6. doi: 10.1016/j.arthro.2005.08.020. PMID 16325083
- [Background] Akasaka T, Nishida J, Imaeda T, Shimamura T, Amadio PC, An KN. Effect of hyaluronic acid on the excursion resistance of tendon graft: a biomechanical in vitro study in a modified human model. Clin Biomech (Bristol). 2006 Oct;21(8):810-5. doi: 10.1016/j.clinbiomech.2006.04.007. Epub 2006 Jun 9. PMID 16762465
- [Background] Akasaka T, Nishida J, Araki S, Shimamura T, Amadio PC, An KN. Hyaluronic acid diminishes the resistance to excursion after flexor tendon repair: an in vitro biomechanical study. J Biomech. 2005 Mar;38(3):503-7. doi: 10.1016/j.jbiomech.2004.04.021. PMID 15652548
- [Background] Nishida J, Araki S, Akasaka T, Toba T, Shimamura T, Amadio PC, An KN. Effect of hyaluronic acid on the excursion resistance of tendon grafts. A biomechanical study in a canine model in vitro. J Bone Joint Surg Br. 2004 Aug;86(6):918-24. doi: 10.1302/0301-620x.86b6.14329. PMID 15330037
- [Background] Hagberg L, Gerdin B. Sodium hyaluronate as an adjunct in adhesion prevention after flexor tendon surgery in rabbits. J Hand Surg Am. 1992 Sep;17(5):935-41. doi: 10.1016/0363-5023(92)90474-4. PMID 1401812
- [Background] Bedi HS, Jowett C, Ristanis S, Docking S, Cook J. Plantaris Excision and Ventral Paratendinous Scraping for Achilles Tendinopathy in an Athletic Population. Foot Ankle Int. 2016 Apr;37(4):386-93. doi: 10.1177/1071100715619989. Epub 2015 Dec 4. PMID 26637273
- [Background] van Schie HT, de Vos RJ, de Jonge S, Bakker EM, Heijboer MP, Verhaar JA, Tol JL, Weinans H. Ultrasonographic tissue characterisation of human Achilles tendons: quantification of tendon structure through a novel non-invasive approach. Br J Sports Med. 2010 Dec;44(16):1153-9. doi: 10.1136/bjsm.2009.061010. Epub 2009 Aug 6. PMID 19666626
- [Background] Docking SI, Rosengarten SD, Cook J. Achilles tendon structure improves on UTC imaging over a 5-month pre-season in elite Australian football players. Scand J Med Sci Sports. 2016 May;26(5):557-63. doi: 10.1111/sms.12469. Epub 2015 May 5. PMID 25943892
- [Background] Docking SI, Rosengarten SD, Daffy J, Cook J. Structural integrity is decreased in both Achilles tendons in people with unilateral Achilles tendinopathy. J Sci Med Sport. 2015 Jul;18(4):383-7. doi: 10.1016/j.jsams.2014.06.004. Epub 2014 Jun 20. PMID 25024134
- [Background] Rosengarten SD, Cook JL, Bryant AL, Cordy JT, Daffy J, Docking SI. Australian football players' Achilles tendons respond to game loads within 2 days: an ultrasound tissue characterisation (UTC) study. Br J Sports Med. 2015 Feb;49(3):183-7. doi: 10.1136/bjsports-2013-092713. Epub 2014 Apr 15. PMID 24735840
- [Background] Pearce CJ, Carmichael J, Calder JD. Achilles tendinoscopy and plantaris tendon release and division in the treatment of non-insertional Achilles tendinopathy. Foot Ankle Surg. 2012 Jun;18(2):124-7. doi: 10.1016/j.fas.2011.04.008. Epub 2011 May 26. PMID 22444000
- [Background] Weinberg EP, Adams MJ, Hollenberg GM. Color Doppler sonography of patellar tendinosis. AJR Am J Roentgenol. 1998 Sep;171(3):743-4. doi: 10.2214/ajr.171.3.9725308. No abstract available.
- [Background] Alfredson H. Midportion Achilles tendinosis and the plantaris tendon. Br J Sports Med. 2011 Oct;45(13):1023-5. doi: 10.1136/bjsports-2011-090217. Epub 2011 May 31. PMID 21628352
- [Background] Calder JD, Freeman R, Pollock N. Plantaris excision in the treatment of non-insertional Achilles tendinopathy in elite athletes. Br J Sports Med. 2015 Dec;49(23):1532-4. doi: 10.1136/bjsports-2014-093827. Epub 2014 Nov 13. PMID 25394422
- [Background] Masci L, Spang C, van Schie HT, Alfredson H. Achilles tendinopathy-do plantaris tendon removal and Achilles tendon scraping improve tendon structure? A prospective study using ultrasound tissue characterisation. BMJ Open Sport Exerc Med. 2015 May 2;1(1):e000005. doi: 10.1136/bmjsem-2015-000005. eCollection 2015. PMID 27900118
- [Background] Robinson JM, Cook JL, Purdam C, Visentini PJ, Ross J, Maffulli N, Taunton JE, Khan KM; Victorian Institute Of Sport Tendon Study Group. The VISA-A questionnaire: a valid and reliable index of the clinical severity of Achilles tendinopathy. Br J Sports Med. 2001 Oct;35(5):335-41. doi: 10.1136/bjsm.35.5.335. PMID 11579069
- [Background] Lintz F, Higgs A, Millett M, Barton T, Raghuvanshi M, Adams MA, Winson IG. The role of Plantaris Longus in Achilles tendinopathy: a biomechanical study. Foot Ankle Surg. 2011 Dec;17(4):252-5. doi: 10.1016/j.fas.2010.08.004. Epub 2010 Sep 15. PMID 22017896
- [Background] Khan KM, Forster BB, Robinson J, Cheong Y, Louis L, Maclean L, Taunton JE. Are ultrasound and magnetic resonance imaging of value in assessment of Achilles tendon disorders? A two year prospective study. Br J Sports Med. 2003 Apr;37(2):149-53. doi: 10.1136/bjsm.37.2.149. PMID 12663358
- [Background] Astrom M, Gentz CF, Nilsson P, Rausing A, Sjoberg S, Westlin N. Imaging in chronic achilles tendinopathy: a comparison of ultrasonography, magnetic resonance imaging and surgical findings in 27 histologically verified cases. Skeletal Radiol. 1996 Oct;25(7):615-20. doi: 10.1007/s002560050146. PMID 8915043
- [Background] McAuliffe S, McCreesh K, Culloty F, Purtill H, O'Sullivan K. Can ultrasound imaging predict the development of Achilles and patellar tendinopathy? A systematic review and meta-analysis. Br J Sports Med. 2016 Dec;50(24):1516-1523. doi: 10.1136/bjsports-2016-096288. Epub 2016 Sep 15. PMID 27633025
- [Background] de Vos RJ, Weir A, van Schie HT, Bierma-Zeinstra SM, Verhaar JA, Weinans H, Tol JL. Platelet-rich plasma injection for chronic Achilles tendinopathy: a randomized controlled trial. JAMA. 2010 Jan 13;303(2):144-9. doi: 10.1001/jama.2009.1986. PMID 20068208
- [Background] Alfredson H, Ohberg L. Sclerosing injections to areas of neo-vascularisation reduce pain in chronic Achilles tendinopathy: a double-blind randomised controlled trial. Knee Surg Sports Traumatol Arthrosc. 2005 May;13(4):338-44. doi: 10.1007/s00167-004-0585-6. Epub 2005 Feb 2. PMID 15688235
- [Background] Chan O, O'Dowd D, Padhiar N, Morrissey D, King J, Jalan R, Maffulli N, Crisp T. High volume image guided injections in chronic Achilles tendinopathy. Disabil Rehabil. 2008;30(20-22):1697-708. doi: 10.1080/09638280701788225. PMID 18608362
- [Background] Wheeler PC, Mahadevan D, Bhatt R, Bhatia M. A Comparison of Two Different High-Volume Image-Guided Injection Procedures for Patients With Chronic Noninsertional Achilles Tendinopathy: A Pragmatic Retrospective Cohort Study. J Foot Ankle Surg. 2016 Sep-Oct;55(5):976-9. doi: 10.1053/j.jfas.2016.04.017. Epub 2016 Jun 7. PMID 27286927
- [Background] Alfredson H, Pietila T, Jonsson P, Lorentzon R. Heavy-load eccentric calf muscle training for the treatment of chronic Achilles tendinosis. Am J Sports Med. 1998 May-Jun;26(3):360-6. doi: 10.1177/03635465980260030301. PMID 9617396
- [Background] Roche AJ, Calder JD. Achilles tendinopathy: A review of the current concepts of treatment. Bone Joint J. 2013 Oct;95-B(10):1299-307. doi: 10.1302/0301-620X.95B10.31881. PMID 24078523
- [Background] Saxena A, Ramdath S Jr, O'Halloran P, Gerdesmeyer L, Gollwitzer H. Extra-corporeal pulsed-activated therapy ("EPAT" sound wave) for Achilles tendinopathy: a prospective study. J Foot Ankle Surg. 2011 May-Jun;50(3):315-9. doi: 10.1053/j.jfas.2011.01.003. Epub 2011 Mar 15. PMID 21406328
- [Background] Lynen N, De Vroey T, Spiegel I, Van Ongeval F, Hendrickx NJ, Stassijns G. Comparison of Peritendinous Hyaluronan Injections Versus Extracorporeal Shock Wave Therapy in the Treatment of Painful Achilles' Tendinopathy: A Randomized Clinical Efficacy and Safety Study. Arch Phys Med Rehabil. 2017 Jan;98(1):64-71. doi: 10.1016/j.apmr.2016.08.470. Epub 2016 Sep 14. PMID 27639439
- [Result] Daseler EH, Anson BJ. The Plantaris muscle an anatomical study of 750 specimens. J Bone Joint Surg [Am] 1943;25-A:822-827.